CLINICAL TRIAL: NCT05064319
Title: Gabapentin for Restoring GABA/Glutamate Homeostasis in Co-occurring Bipolar and Cannabis Use Disorders: A Randomized, Double-blind, Placebo-controlled, Parallel-group, MRI Study
Brief Title: Gabapentin for Restoring GABA/Glutamate Homeostasis in Co-occurring Bipolar and Cannabis Use Disorders
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, James Prisciandaro, Associate Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00112593; R01DA054275 (NIH)
Record Dates: First submitted 2021-09-22; First posted 2021-10-01 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Bipolar Disorder; Cannabis Use; Schizoaffective Disorder, Bipolar Type; Bipolar I Disorder; Bipolar II Disorder; Cannabis Use Disorder, Mild; Cannabis Use Disorder, Moderate; Cannabis Use Disorder, Severe
MeSH Terms: conditions — Bipolar Disorder; Psychotic Disorders; Lymphoma, Follicular | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A - Gabapentin (Experimental)
  Interventions: Drug: Gabapentin
- Group B - Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — After group assignment but before taking any study medication, and again 17 days later, participants will have a Magnetic Resonance Imaging (MRI) exam after completing various assessments (clinical interview, questionnaires, etc.). Group A will receive gabapentin 2-3 times a day for a total of 17 days.
  Arms: Group A - Gabapentin
Drug: Placebo — After group assignment but before taking any study medication, and again 17 days later, participants will have a Magnetic Resonance Imaging (MRI) exam after completing various assessments (clinical interview, questionnaires, etc.). Group A will receive placebo 2-3 times a day for a total of 17 days.
  Arms: Group B - Placebo

SUMMARY:
This research study evaluates the effects of an FDA-approved medication Gabapentin in individuals with Bipolar Disorder who smoke marijuana. Participants in the study will will be assigned to take either Gabapentin or a matched placebo. Study medication will be taken for 17 days. There will be 5 study visits, with 2 MRI brain imaging scans completed. Questionnaires and clinical interview measures will be completed at study visits along with consistent assessment of potential side effects from study medication.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-65 years
2. Meet DSM-5 criteria for moderate or severe cannabis use disorder (CUD; within the past 3 months), provide a positive urine cannabinoid screen at baseline, and identify cannabis as the primary substance of abuse
3. Meet DSM-5 criteria for bipolar I or II disorder (BD) or Schizoaffective Disorder, Bipolar Type
4. Able to provide informed consent and read, understand, and accurately complete assessment instruments
5. Willing to commit to medication treatment and follow-up assessments
6. Prescribed daily use of at least one mood stabilizing medication (i.e., lithium, divalproex sodium, lamotrigine, carbamazepine, 2nd generation antipsychotic)

Exclusion Criteria:

1. A primary psychiatric diagnosis other than BD (e.g., Schizophrenia)
2. Meet DSM-5 criteria for moderate or severe substance use disorder (other than cannabis or tobacco) within the past 60 days
3. Any uncontrolled neurological condition (e.g., epilepsy) that could confound the results of the study
4. Any history of brain injury with loss of consciousness greater than 5 minutes
5. Any history of mental retardation, dementia, or recent electroconvulsive therapy (in the past 3 months)
6. Any uncontrolled medical condition that may adversely affect the conduct of the study or jeopardize the safety of the participant
7. Hepatocellular disease as indicated by plasma levels of liver transaminases (aspartate transaminase, alanine transaminase) greater than 3 times the normal range
8. Renal insufficiency as indicated by plasma levels of creatinine greater than 2 times the normal range
9. Concomitant use of medications that could interfere with glutamatergic/GABAergic transmission (e.g., benzodiazepines, ceftriaxone, riluzole, memantine, ketamine, topiramate, vigabatrin), due to potential confounding effects
10. Concomitant use of opioid medications, benzodiazepines, barbiturates, chloral hydrate, sodium oxybate, or any other medication deemed to be hazardous if taken with gabapentin
11. Azelastine, orphenadrine, oxomemazine, paraldehyde, and thalidomide are generally contraindicated in patients taking gabapentin; as such, individuals taking these medications will be excluded
12. Women of childbearing potential who are pregnant, lactating, or refuse adequate forms of contraception
13. Current suicidal or homicidal risk
14. Baseline scores greater than 35 on the Montgomery-Asberg Depression Rating Scale or greater than 25 on the Young Mania Rating Scale
15. Has taken gabapentin in the last month or experienced adverse effects/allergic reaction (e.g., angioedema) from it at any time
16. Significant claustrophobia and/or past negative experiences with MRI
17. Presence of non-MRI safe materials in the body (e.g., ferrous metal implants, pacemaker)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-02-24 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in prefrontal GABA concentrations through Proton Magnetic Resonance Spectroscopy | Baseline to end of treatment, approximately 17 days
  Concentrations of GABA, normalized to water and corrected for CSF%, in dorsal anterior cingulate measured via Proton Magnetic Resonance Spectroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: James J Prisciandaro, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University Of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No